CLINICAL TRIAL: NCT01853930
Title: Translation of Eye Movement Reading Training to Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C0849-R
Record Dates: First submitted 2013-05-02; First posted 2013-05-15 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Macular Disease
Keywords: reading rehabilitation; macular degeneration; eccentric viewing
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laboratory training (Other): Patients will be trained in the laboratory with feedback by a rehabilitation therapist
  Interventions: Behavioral: Platform for Administering Eye-movement Control Training
- Home-based training (Other): Patients will self instruct using the computer-based training with remote intervention by a therapist
  Interventions: Behavioral: Platform for Administering Eye-movement Control Training

INTERVENTIONS:
Behavioral: Platform for Administering Eye-movement Control Training — The Platform for Administering Eye-movement Control Training (PAECT) meta program will incorporate all of the exercises that the investigators have developed and validated over the course of our previous Merit Review grants (Seiple, Szlyk et al., 2005, 2011). The PAECT platform will be designed to allow patients to easily run the training exercises in their homes and to practice at their convenience. The PAECT will employ an executive component that will keep track of the exercises that are practiced and record performance. Each time a subject opens the platform, it will choose the exercise for that subject based upon previous training and performance.

SUMMARY:
Age-related macular degeneration (AMD) is the most common visual impairment in persons over 50 years of age. It has been estimated that 1 in 3 individuals over 75 years of age and 1 in 30 individuals over 52 years of age are affected by AMD. The deficits in visual function as a result of this disease affecting the central retina are debilitating, as individuals lose their ability to carry out many of their daily activities that require resolving fine spatial details. The investigator's previous studies have shown that training with oculomotor control exercises significantly increases reading speeds in patients with AMD. In the proposed study, the investigators will examine whether these training exercises are effective when practiced at home.

In Phase 1, the investigators will develop a standardized user-friendly, Web-based platform that will allow patients to easily self-administer training exercises. The software platform will be designed to automatically choose the appropriate exercises based on a patient's previous performance, run the training exercise, and collect performance data into a universal patient data file. In Phase 2, the platform will be tested in two settings: in standard clinical rehabilitation practice and in the patient's home. Reading outcomes in the two settings will be compared. The investigators will recruit 60 patients per year for each of the three years for Phase 2 of the study. Half of these patients will be assigned to the Clinic Training Group, while the other half will be assigned to At-home Training Group. For all patients, three assessments will be taken: at baseline, after 1 month, and after 2 months of training.

The investigators will compare reading outcomes to assess the roles of feedback versus the role of frequent available practice. Because of the extensive cost and clinical resources required for vision rehabilitation, it is critical to determine whether the training program can be made less expensive, but as effective, when it is self-trained. If the investigators demonstrate the utility of at-home practice, clinical facilities and therapists' time can be made available for those activities requiring face-to-face contact

DETAILED DESCRIPTION:
In the proposed study, the investigators will examine whether these training exercises are effective when practiced at home. There are two specific aims in this project:

Aim #1 (Year 1): to develop a web-based meta program that will administer the training exercises. For convenience, in this proposal, the investigators will refer to this platform as PAECT (Platform for Administering Eye movement Control Training). The PAECT meta program will incorporate all of the exercises that the investigators have developed and validated over the course of our previous Merit Review grants (Seiple, Szlyk et al., 2005, 2011). The PAECT platform will be designed to allow patients to easily run the training exercises in their homes and to practice at their convenience. The PAECT will employ an executive component that will keep track of the exercises that are practiced and record performance. Each time a subject opens the platform, it will choose the exercise for that subject based upon previous training and performance. The development of the software and the design of the hardware interface for administering the system will take place during the first year of the project. This will be done through a series of software/hardware iterations based upon feedback derived from direct patient testing of the system. The investigators will recruit ten patients with AMD to test and comment on the system during this phase of the project.

Aim #2 (Years 2-4). To compare the effects of PAECT training on reading outcomes in two training situations: (1). training done in the clinic with feedback on performance provided by a trained low-vision therapist, and (2) training done at-home with expanded opportunity for practicing the exercises, but with no therapist feedback. Patients will be assigned to one of two groups: Patients in Group 1 ("Clinical") will undergo weekly two-hour training sessions for three months using the software/hardware system. This training will be conducted in the low-vision clinic using the PAECT, with feedback on performance provided by a trained low-vision therapist. Patients in Group 2 ("At-home") will practice all of the exercises at home using the PAECT system over a three-month period. The subjects will be encouraged to use the system as often as possible, but no less than two hours per week. Sixty patients (30 in the clinical setting and 30 at home) will be tested for each of three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of retinal disease affecting the central visual field (e.g., non-exudative "dry" AMD)
* with a central scotoma
* and with visual acuity of less than or equal to 20/70 and greater than or equal to 20/400 (in the test eye), will be included in the study.
* The presence of a central scotoma and eccentric viewing will be confirmed using an OPKO OCT/SLO microperimetry.
* The investigator's intent is to include subjects based upon the patient's functional characteristics (e.g., eccentric viewing).

Exclusion Criteria:

* Patients with other major ophthalmologic or neurologic disease
* choroidal neovascularization ("wet" AMD)
* moderate to severe media opacities
* and cognitive impairment will be excluded.
* Patients' disease status will be monitored throughout the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet P Szlyk, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ming J, Thulborn KR, Szlyk JP. Reproducibility of activation maps for longitudinal studies of visual function by functional magnetic resonance imaging. Invest Ophthalmol Vis Sci. 2012 Sep 14;53(10):6153-63. doi: 10.1167/iovs.11-8375. PMID 22879425
- [Result] Grant P, Seiple W, Szlyk JP. Effect of depression on actual and perceived effects of reading rehabilitation for people with central vision loss. J Rehabil Res Dev. 2011;48(9):1101-8. doi: 10.1682/jrrd.2010.05.0080. PMID 22234714
- [Result] Seiple W, Grant P, Szlyk JP. Reading rehabilitation of individuals with AMD: relative effectiveness of training approaches. Invest Ophthalmol Vis Sci. 2011 May 5;52(6):2938-44. doi: 10.1167/iovs.10-6137. PMID 21296824
- [Result] Szlyk JP, Little DM. An FMRI study of word-level recognition and processing in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2009 Sep;50(9):4487-95. doi: 10.1167/iovs.08-2258. Epub 2009 Apr 22. PMID 19387076
- [Result] Soong GP, Shapiro M, Seiple W, Szlyk JP. Macular structure and vision of patients with macular heterotopia secondary to retinopathy of prematurity. Retina. 2008 Oct;28(8):1111-6. doi: 10.1097/IAE.0b013e3181744136. PMID 18779718
- [Result] Little DM, Thulborn KR, Szlyk JP. An FMRI study of saccadic and smooth-pursuit eye movement control in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2008 Apr;49(4):1728-35. doi: 10.1167/iovs.07-0372. PMID 18385097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 patients were screened for eligibility between January 2014 and June 2017 at the Jesse Brown VA Medical Center in Chicago, Illinois.
Pre-assignment Details: 33 patients were assigned to either the laboratory training group or the home-based training group. 14 were assigned to the focus group during the developmental phase (year 1) of the web-based meta program and are not included in the analysis of outcome measures. 26 did not meet the inclusion criteria and 25 declined to participate.
Groups:
- Laboratory Training: Patients will be trained in the laboratory by a rehabilitation therapist
  The Platform for Administering Eye movement Control Training (PAECT) meta program will incorporate all of the exercises that the investigators have developed and validated over the course of our previous Merit Review grants (Seiple, Szlyk et al., 2005, 2011). The PAECT platform will be designed to allow future patients to easily run the training exercises in their homes and to practice at their convenience. The PAECT will employ an executive component that will keep track of the exercises that are practiced and record performance. Each time a subject opens the platform, it will choose the exercise for that subject based upon previous training and performance.
- Home-based Training: Patients will self instruct using the computer-based training with remote intervention by a therapist as needed
  The Platform for Administering Eye movement Control Training (PAECT) meta program will incorporate all of the exercises that the investigators have developed and validated over the course of our previous Merit Review grants (Seiple, Szlyk et al., 2005, 2011). The PAECT platform will be designed to allow future patients to easily run the training exercises in their homes and to practice at their convenience. The PAECT will employ an executive component that will keep track of the exercises that are practiced and record performance. Each time a subject opens the platform, it will choose the exercise for that subject based upon previous training and performance.
Period: Overall Study
Arm/Group | Laboratory Training | Home-based Training
Started | 25 | 8
Completed | 25 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laboratory Training | Home-based Training | Total
Number analyzed (Participants) | 25 | 8 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 2 | 13
  >=65 years | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (24.1) | 75.9 (11.9) | 68.1 (22.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 21
  Male | 9 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 17 | 7 | 24
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 8 | 33
Reading Performance and Accuracy [Mean (Standard Deviation); unit: Words Per Minute (WPM)] | 60.4 (41.1) | 40.9 (35.6) | 55.7 (40.2)
Visual Acuity [Mean (Standard Deviation); unit: logMAR] | 0.95 (0.23) | 0.98 (0.27) | 0.96 (0.24)
Contrast [Mean (Standard Deviation); unit: logCS] | 1.01 (0.43) | 1.08 (0.41) | 1.03 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Change in Reading Performance and Accuracy Using MNREAD.
Description: Participants will be trained to use eccentric viewing for reading. They will then be assessed on the following outcome measures; reading, speed and accuracy using the MNRead test, binocular visual acuity and contrast sensitivity.
Time Frame: Participants will be assessed at baseline, 1 month and 2 months but change between baseline and final (2 months) will be reported
Population: All 33 participants who received and completed training on the PAECT platform for eight weeks (in the laboratory or at-home) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Words Per Minuted (WPM)
Arm/Group | Laboratory Training | Home-based Training
Number analyzed (Participants) | 25 | 8
Words Per Minuted (WPM) | 22.59 (26.51) | 24.68 (17.76)
Statistical Analysis 1: Comparison: Laboratory Training vs Home-based Training; Test type: Superiority — The purpose of the superiority test is to show if laboratory based training is superior to an independent home-based training option; p = 0.876, t-test, 2 sided; t= -0.157 df= 30

ADVERSE EVENTS:
Time Frame: Participants were assessed at baseline, 1 month and 2 months.
Arm/Group | Laboratory Training | Home-based Training
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/8
Other Adverse Events (participants affected / at risk) | 0/25 | 0/8

LIMITATIONS AND CAVEATS:
Future research will address some of the limitations of this study such as greater diversity of subjects, a larger sample size and additional development and refinement of the program interface and user experience.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT01853930/Prot_SAP_000.pdf